CLINICAL TRIAL: NCT00140374
Title: Phase I/II Study of Vaccination Priming and Vaccine Boosting With Allogeneic Human GM-CSF Gene Transduced Irradiated Prostate Cancer Cell Vaccines in Patients With Prostate Cancer
Brief Title: Vaccination Priming and Vaccine Boosting Trial of Allogeneic Human GM-CSF Gene Transduced Irradiated Prostate Cancer Cell Vaccines (GVAX® Vaccine for Prostate Cancer)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Genesys (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-9705A
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2005-09-01 (Estimated); Status verified 2005-08

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Vaccine; GVAX; Allogeneic cells
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

INTERVENTIONS:
Biological: Immunotherapy allogeneic GM-CSF secreting cellular vaccine

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of priming vaccinations, and subsequent boosting vaccinations with GVAX® Vaccine for Prostate Cancer. Clinical observations and laboratory measurements will be monitored to evaluate safety and toxicity. Additionally, the antitumor effects of GVAX® Vaccine for Prostate Cancer on serum PSA levels, will be evaluated and antitumor responses will be quantitated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma prostate cancer that has recurred after surgery by PSA
* No evidence of measurable metastatic disease
* An ECOG performance status of 0 or 1

Exclusion Criteria:

* Transitional cell, small cell or squamous cell prostate carcinomas
* Any previous radiation therapy, prior anti-androgens or prior investigational therapy
* Previous hormonal therapy of any type for prostate cancer
* Previous biological therapy for cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 1998-12; Study Completion 2001-02